CLINICAL TRIAL: NCT02827422
Title: A Prospective, Multicenter Registry With Targeted Temperature Management After Out-of-hospital Cardiac Arrest in Korea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kyu Nam Park (Other)
Responsible Party: Sponsor-Investigator, Kyu Nam Park, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: 2015-P33001-00
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: therapeutic hypothermia
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: not provided

SUMMARY:
Therapeutic hypothermia after out-of-hospital cardiac arrest is considered as a standard care. However, optimal candidates, optimal dose, duration, timing of initiation and rate of rewarming is still unknown. The objective of this project is to improve the outcomes for patients after resuscitation from out-of-hospital cardiac arrest treated with therapeutic hypothermia established from the analysis of multicenter registry data.

ELIGIBILITY:
Inclusion Criteria:

* age of older than 18 years
* out-of-hospital cardiac arrest
* comatose mentality after return of spontaneous circulation (ROSC)
* treated with therapeutic hypothermia, regardless of target temperature

Exclusion Criteria:

* suspected or confirmed to cerebrovascular accident
* poor pre-arrest neurologic status (CPC>3)
* patients who are terminally ill or for whom intensive care dose not seem to be appropriate
* Do not attempt resuscitation (DNAR) order
* patients with tympanic membrane temperature below 30 degree celsius on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with therapeutic hypothermia after out-of-hospital cardiac arrest.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
survival | 6 months after cardiac arrest
Neurologic Outcome | 6 months after cardiac arrest
  Cerebral Performance Category (CPC). CPC 1,2 : Good Outcome CPC 3,4,5 : Poor Outcome
Neurologic Outcome | after 6 months
  modified Rankin Scale (mRS) mRS 0,1,2, 3 : Good Outcome mRS 4,5,6 : Poor Outcome

SECONDARY OUTCOMES:
survival | duration of hospitalization, limit 180 days
neurological outcome | duration of hospitalization, limit 180 days
  Cerebral Performance Category (CPC). CPC 1,2 : Good Outcome CPC 3,4,5 : Poor Outcome
neurological outcome | duration of hospitalization, limit 180 days
  modified Rankin Scale (mRS) mRS 0,1,2, 3 : Good Outcome mRS 4,5,6 : Poor Outcome
Survival | 1 month after cardiac arrest
neurological outcome | 1 month after cardiac arrest
  Cerebral Performance Category (CPC). CPC 1,2 : Good Outcome CPC 3,4,5 : Poor Outcome
neurological outcome | 1 month after cardiac arrest
  modified Rankin Scale (mRS) mRS 0,1,2, 3 : Good Outcome mRS 4,5,6 : Poor Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Nam Park, MD. PhD, Principal Investigator — Seoul St. Mary's Hospital, The Catholic University of Korea
Locations (1):
- Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim YJ, Kim YH, Youn CS, Cho IS, Kim SJ, Wee JH, Park YS, Oh JS, Lee BK, Kim WY. Different neuroprognostication thresholds of neuron-specific enolase in shockable and non-shockable out-of-hospital cardiac arrest: a prospective multicenter observational study in Korea (the KORHN-PRO registry). Crit Care. 2023 Aug 9;27(1):313. doi: 10.1186/s13054-023-04603-6. PMID 37559163
- [Derived] Oh JH, Lee DH, Cho IS, Youn CS, Lee BK, Wee JH, Cha KC, Chae MK, Shin J; Korean Hypothermia Network Investigators. Association between acute kidney injury and neurological outcome or death at 6 months in out-of-hospital cardiac arrest: A prospective, multicenter, observational cohort study. J Crit Care. 2019 Dec;54:197-204. doi: 10.1016/j.jcrc.2019.08.029. Epub 2019 Aug 28. PMID 31521016